CLINICAL TRIAL: NCT05461066
Title: Tobacco Cessation Care Service in the Community Pharmacy: Cost-effectiveness of a Non-randomized Cluster-controlled Trial at 12-months' Follow-up
Brief Title: Cost-effectiveness of a Tobacco Cessation Care Service in the Community Pharmacy
Acronym: CESAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Espanola de Farmacia Clinica, Familiar y Comunitaria (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EPA-13-16
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Smoking Cessation; Pharmacist-Patient Relations
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Smoking cessation intervention in community pharmacies
  Interventions: Behavioral: CESAR training
- Control (Active Comparator): Usual care of smoking cessation in community pharmacies
  Interventions: Behavioral: CESAR training

INTERVENTIONS:
Behavioral: CESAR training — Intervention community pharmacists received the CESAR training to improve their smoking cessation services, consisting of an initial interview and follow-up visits to identify obstacles and reinforce behaviours.

SUMMARY:
The study was a non-randomized controlled trial of 12-months' follow-up with 182 Spanish community pharmacists. Intervention community pharmacists received the CESAR training to improve their smoking cessation services, consisting of an initial interview and follow-up visits to identify obstacles and reinforce behaviours. The control group received the usual care. Data were self-reported and collected in a computerized health registration system. Outcomes were smoking cessation and quality of life (EuroQOL-5D) collected at baseline, 6 months', and 12 months' follow-up. Cost data were collected for the study period and included direct health costs, sick leave, and intervention costs. Smoking cessation was analysed through logistic regression models. Generalized linear models were carried out for quality-adjusted life year costs. Incremental cost-effectiveness ratios (ICERs) and cost-utility ratios (RCUI) were calculated. Sensitivity analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

* smoker over 18 years old
* consent to participate
* presence at the community pharmacy for one of three reasons (a) a medical prescription for a treatment to stop smoking, (b) a consultation about how to stop smoking, (c) asking if he/she smokes when he/she consults for associated symptoms or harm.

Exclusion Criteria:

* cognitive impairment
* drug uses
* pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | Before/after the intervention (1 year)
  Dichotomicus variable (yes/no)
Quality of Life (EuroQOL-5D) | 1 year
  Measured with EuroQOL-5D
Cost-effectiveness | 1 year
  In cost-effectiveness, the deterministic Incremental Cost Effectiveness Ratio (ICER) is the coefficient resulting from dividing the difference between groups in costs by the difference in probability between groups that an additional patient will cease their smoking history.
Cost-utility | 1 year
  For the cost-utility, the Deterministic Incremental Cost-Utility Ratio (ICUR) is the coefficient resulting from dividing the difference between groups in costs by the difference between groups in quality-adjusted life years.

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Gomez Martinez JC, Gaztelurrutia Lavesa L, Mendoza Barbero A, Plaza Zamora J, Lage Pinon M, Aguilo Juanola M, Climent Catala M, de Andres Dirube A, Garcia Moreno L, Jaraiz Magarinos I, Moral Ajado M, Sanchez Marcos N. Smoking cessation intervention in the community pharmacy: Cost-effectiveness of a non-randomized cluster-controlled trial at 12-months' follow-up. Res Social Adm Pharm. 2024 Jan;20(1):19-27. doi: 10.1016/j.sapharm.2023.09.003. Epub 2023 Sep 7. PMID 37704533